CLINICAL TRIAL: NCT05938088
Title: Mirogabalin and Pain After Total Hip Arthroplasty: a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Mirogabalin for Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Do-Hyeong Kim, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3-2023-0151
Record Dates: First submitted 2023-06-29; First posted 2023-07-10 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mirogabalin group (Experimental): perioperative mirogabalin
  Interventions: Drug: Arm I (mirogabalin group)
- placebo group (Sham Comparator): placebo
  Interventions: Drug: Arm II (placebo group)

INTERVENTIONS:
Drug: Arm I (mirogabalin group) — Take two capsules of Mirogabalin 5 mg within 30 minutes before going to the operating room. Patients take 5 mg of mirogabalin twice daily at 12-hour intervals until POD 7 days.
  Arms: mirogabalin group
Drug: Arm II (placebo group) — It is performed in the same way as Arm l.
  Arms: placebo group

SUMMARY:
The purpose of this study is to confirm the analgesic effect of mirogabalin in patients undergoing unilateral hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 19 years of age or older who are expected to undergo unilateral hip arthroplasty
2. American Society of Anesthesiologists class 1-3

Exclusion Criteria:

1. Major prior ipsilateral open hip surgery
2. Allergies to drugs used in research
3. Difficult to manage diabetes mellitus (including insulin dependence)
4. Chronic use of gabapentin or pregabalin (regular use for more than 3 months)
5. Patients taking cimetidine, probenecid, or lorazepam
6. Patients with moderate or severe hepatic impairment (AST/ALT 2.5 times or more of the upper limit of normal)
7. Estimated glomerular filtration rate < 60 mL/min/1.73m2
8. Dependence on opioids
9. In the case of subjects who cannot read the consent form (e.g. illiterate, foreigners, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-06-28 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
numeric rating scale at flexion | postoperative day 1
  A score of 0 indicates no pain and a score of 10 indicates maximum pain.

SECONDARY OUTCOMES:
numeric rating scale at flexion | up to 3 month after surgery
  A score of 0 indicates no pain and a score of 10 indicates maximum pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea